CLINICAL TRIAL: NCT07013656
Title: Effects of Combined Intraduodenal Administration of Calcium and L-tryptophan on Plasma Glucose, Glucoregulatory Hormones and Gastric Emptying in Response to a Mixed-nutrient Drink in Healthy Adult Males
Brief Title: Effects of Combined Administration of Calcium and L-tryptophan on Gut Functions and Blood Glucose in Healthy Humans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Christine Feinle-Bisset, Professor Christine Feinle-Bisset (Professorial Senior Research Fellow), University of Adelaide
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 13243
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Intraduodenal; Calcium; L-tryptophan; Gastric emptying; Glucoregulatory hormones; Plasma glucose; Human
MeSH Terms: interventions — Tryptophan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- L-tryptophan (Active Comparator): In this arm, participants will receive a 75-minute intraduodenal infusion of an isotonic solution containing 1.83 g L-tryptophan, dissolved in 225 mL distilled water. Additionally, 2.2 g of sodium chloride (NaCl) will be added to ensure the solution is isosmotic (~373 mOsm).
  Interventions: Other: L-tryptophan
- L-tryptophan + Ca-500 (Active Comparator): In this arm, participants will receive a 75-minute intraduodenal infusion of an isotonic solution containing 1.83 g L-tryptophan and 1.84 g of calcium chloride dihydrate (CaCl₂·2H₂O), dissolved in 225 mL of distilled water. Additionally, 1.1 g of NaCl will be added to ensure the solution is isosmotic (~373 mOsm).
  Interventions: Other: Combination of L-tryptophan + Ca-500
- L-tryptophan + Ca-1000 (Active Comparator): In this arm, participants will receive a 75-minute intraduodenal infusion of an isotonic solution containing 1.83 g L-tryptophan and 3.68 g of calcium chloride dihydrate (CaCl₂·2H₂O), dissolved in 225 mL of distilled water. This solution has an osmolality of ~373 mOsm.
  Interventions: Other: Combination of L-tryptophan + Ca-1000
- Control (Placebo Comparator): In this arm, participants will receive a 75-minute intraduodenal infusion of saline (an isotonic solution containing 2.5 g of NaCl, dissolved in 225 mL of distilled water). This solution has an osmolality of ~373 mOsm.
  Interventions: Other: Control

INTERVENTIONS:
Other: L-tryptophan — L-tryptophan, an aromatic amino acid and one of the building blocks of protein, is a part of our daily diet. The load of L-tryptophan (0.1 kcal/minute) is based on our previous study, in which L-tryptophan represented a submaximal load.
  Arms: L-tryptophan
Other: Combination of L-tryptophan + Ca-500 — Calcium, an essential mineral and a key component of dairy products, is a regular part of our daily diet. In this condition, both L-tryptophan and calcium will be administered as 'active'. Recent studies have shown that calcium in a dose of 500 mg enhances the effects of L-tryptophan to stimulate gut functions and reduce energy intake. This dose of calcium will be considered 'lower dose'.
  Arms: L-tryptophan + Ca-500
Other: Combination of L-tryptophan + Ca-1000 — In this condition, both L-tryptophan and calcium will be administered. In our study calcium in a dose of 1000 mg enhances the effects of L-tryptophan to stimulate gut functions and reduce energy intake. This dose of calcium will be considered 'higher dose'.
  Arms: L-tryptophan + Ca-1000
Other: Control — An isotonic solution containing 2.5 g of NaCl, dissolved in 225 mL of distilled water.
  Arms: Control

SUMMARY:
The intervention in this study consists of 75-minute intraduodenal infusions of isosmotic solutions containing either saline (control), L-tryptophan, or calcium combined with L-tryptophan. Participants enrolled into the study will receive, in a randomised, double-blind fashion either (i) saline (control), (ii) L-tryptophan at a rate of 0.1 kcal/minute, (iii) combination of L-tryptophan (0.1 kcal/minute) + 500 mg calcium, or (iv) combination of L-tryptophan (0.1 kcal/minute) + 1000 mg calcium in four separate sessions, each of which will be separated by at least 4 (and up to 10) days. Each study session will be 4-6 hours. Studies will be carried out in the Clinical Research Facility of the Adelaide Medical School, the University of Adelaide, by staff and students trained in the required techniques.

DETAILED DESCRIPTION:
Each participant will be required to consume a standardised dinner meal (beef lasagne; total energy content: 602 kcal; McCain Food, Wendouree, Victoria, Australia) on the night before each visit by 7 pm. After fasting overnight for ~ 13.5 hours and refraining from exercise and alcohol during the previous 24 hours, the participant will arrive in the laboratory at 8.30 am. After confirming adherence to the study requirements, vital signs ( blood pressure, heart rate and body temperature) will be measured to establish baseline values for safety, and they will be monitored throughout the study. Then, a manometric catheter will be inserted through an anaesthetised nostril and allowed to pass through the stomach and into the duodenum by peristalsis. The infusion port will be positioned ~ 14 cm distal to the pylorus. The correct positioning of the catheter will be monitored continuously by measurement of the transmucosal potential difference in the stomach (~ -40 mV) and the duodenum (~ 0 mV). Once the catheter has been positioned correctly, an intravenous cannula will be placed into a forearm vein for regular blood sampling. At time = -30 minute, a baseline blood sample (6 ml), visual analogue scale (VAS) questionnaire to assess gastrointestinal (GI) symptoms, and breath sample to assess gastric emptying will be collected. Then the infusion of one of the study treatments, i.e. (i) saline, (ii) L-tryptophan, (iii) L-tryptophan + 500 mg calcium, or (iv) L-tryptophan + 1000 mg calcium, will commence and continue for 75 minutes (times = -30 to 45 minutes). At time = -1 minute, participants will consume, within 1 minute, a mixed-nutrient drink (350 mL, containing 500 kcal, 74 g carbohydrates) labelled with 100 mg 13C-acetate for measurement of gastric emptying by non-invasive breath sampling at regular intervals, for subsequent analysis of 13CO2 levels. Blood samples for the measurement of plasma glucose and hormone concentrations, and VAS questionnaires, will be collected before and after the mixed-nutrient drink. At time = 240 minute, after collecting final blood and breath samples and VAS questionnaire, the intravenous cannula will be removed and the participant will be served a light lunch, after which they will be allowed to leave the laboratory. A total of 84 mL of blood (14 sampling time points, 6 mL each) will be taken on each study day (study total of 344 mL, including screening).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, lean males (only men will be included in the study to avoid the confounding effects of the menstrual cycle on gastric emptying).
* BMI: 19-25 kg/m2,
* Weight-stable (i.e. <5% fluctuation) at study entry, which will be ascertained by a stable body weight in the preceding 3 months.

Exclusion Criteria:

* Significant GI symptoms, or history of GI disease or surgery
* Current gallbladder or pancreatic disease
* Cardiovascular or respiratory diseases
* Any other illnesses as assessed by the investigator (including chronic illnesses not explicitly listed above)
* Use of prescribed or non-prescribed medications (including vitamins and herbal supplements) which may affect energy metabolism, GI function, body weight or appetite (e.g. domperidone, cisapride, anticholinergic drugs (e.g. atropine), metoclopramide, erythromycin, hyoscine, orlistat, green tea extracts, Astragalus, St Johns Wort etc.)
* Lactose intolerance/other food allergy(ies)
* Individuals with low ferritin levels (<30 ng/mL), or who have donated blood in the 12 weeks prior to taking part in the study
* High performance athletes
* Current intake of > 2 standard drinks on > 5 days per week (>140g/week)
* Current smokers of tobacco (cigarettes, cigars, pipes, sheesha, chewing, vaping etc.)
* Current use of recreational drugs, e.g. marijuana
* Current intake of any illicit substance
* Vegetarians
* Inability to tolerate nasoduodenal tube
* Inability to comprehend study protocol
* Restrained eaters (score >12 on the 3-factor eating questionnaire)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06-28 (Estimated); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose concentrations | Blood samples will be collected over 4.5 hours: at baseline (time = -30 minutes), then at regular intervals before and after drink administration (times = -25, -15, 0, 10, 20, 30, 45, 60, 75, 90, 120, 180, and 240 minutes).
  Plasma glucose concentrations (mmol/L) will be assessed using the glucose oxidase method.

SECONDARY OUTCOMES:
Gastric emptying | Breath samples will be collected in sealed tubes over 4.5 hours: at baseline (time = -30 minutes), prior to treatment administration, every 5 minutes after the drink (times = 0 to 60 minutes), and then every 10 minutes until 240 minutes post-drink.
  13C-acetate breath test, measuring 13CO2 levels in end-expiratory breath samples.
Plasma concentrations of glucoregulatory hormones e.g. glucagon-like peptide (GLP-1), glucose-dependent insulinotropic polypeptide (GIP), C-peptide, glucagon, insulin and cholecystokinin (CCK) | Blood samples will be collected over 4.5 hours: at baseline (time = -30 minute), then at regular intervals before and after the drink (times = -25, -15, 0, 10, 20, 30, 45, 60, 75, 90, 120, 180, and 240 minutes).
  Plasma concentrations of hormones e.g. GLP-1, GIP and CCK (pmol/L) will be determined using radioimmunoassays, and plasma C-peptide, glucagon and insulin concentrations (pmol/L) will be measured using ELISA immunoassays.
GI symptoms (nausea and bloating) will be assessed as a composite secondary outcome. | VAS questionnaires will be collected over 4.5 hours: at baseline (time = -30 minutes), at regular intervals before and after the drink (times = -15, 0, 10, 20, 30, 45, 60, 75, and 90 minutes), then every 10 minutes until 240 minutes post-drink.
  These will be measured using 100mm VAS questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Christine Feinle-Bisset, Principal Investigator — Adelaide Medical School University of Adelaide Level 5 Adelaide Health and Medical Sciences Building, Cnr George St and North Tce, Adelaide, SA 5005
Locations (1):
- Clinical Research Facility, Adelaide Health and Medical Sciences Building, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
The de-identified individual participant data (IPD) collected during the study will not be shared with other researchers. This is due to the ethical approval and informed consent process, which require that data remain confidential and not be shared outside the primary research group, even in de-identified form.